CLINICAL TRIAL: NCT01066390
Title: A Study on the Safety and Immunogenicity of Combined Intradermal and Intravenous Administration of an Autologous mRNA Electroporated Dendritic Cell Vaccine in Patients With Previously Treated Unresectable Stage III or IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bart Neyns (Other)
Responsible Party: Sponsor-Investigator, Bart Neyns, MD PhD, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-015748-40
Record Dates: First submitted 2010-01-08; First posted 2010-02-10 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2012-08

CONDITIONS: Melanoma
Keywords: stage IIIC/IV melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: TriMix-DC — eligible patients will undergo a leucapheresis for the preparation of autologous TriMix-DC vaccine.4 weeks after the leucapheresis patients will initiate therapeutic vaccination with the TriMix-DC vaccine by IV and ID administration. The vaccines will be administered at 4 different visits that will be separated with an interval of 2 weeks.

SUMMARY:
This phase I study plan is divided in the following four phases:

* Eligibility Screen Phase (week -4 to -1): Following written informed consent patients with metastatic melanoma (AJCC stage III/IV with unresectable disease) will undergo an eligibility screen (incl. blood analysis and PET/CT-scan).
* TriMix-DC Vaccine Manufacturing Phase (week I to IV): eligible patients will undergo a leucapheresis (15 liter of venous blood) for the preparation of autologous TriMix-DC vaccine. Vaccine preparations will be manufactured and quality-controlled (during an interval of 4 weeks following the leucapheresis) and released for patient administration if the TriMix-DC preparation fulfills the predefined quality requirements.
* TriMix-DC Vaccine Administration Phase (Week 1 to 24): 4 weeks after the leucapheresis patients will initiate therapeutic vaccination with the TriMix-DC vaccine by IV and ID administration. The vaccines will be administered at 4 different visits that will be separated with an interval of 2 weeks. At each vaccination a total of 12.106 DC per antigen will be administered.
* Patients will be allocated to three different cohorts:

  * The first cohort will receive 10% of TriMix-DC by iv and 90% by id injection.
  * The second cohort 25% by iv and 75% by id injection.
  * The third cohort 50% by iv and 50% by id injection.
* During the week following the administration of the fourth vaccine (= week 8), a DTH-test and punch biopsy of the injection site will be performed as well as a second leucapheresis (for the purpose of immuno-monitoring) and tumor evaluation (by PET-CT).
* A fifth vaccine will be administered and a repeat tumor staging performed in week 16 (= 8w after the fourth vaccine).
* End of study visit: Patients will perform an "end of study visit" 8 weeks after the fifth vaccine (= week 24) as well as a new tumor evaluation (PET/CT).
* Follow-up Phase: survival data will be obtained until 3 years after the initiation of vaccine therapy or the time of death.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give valid written informed consent before undergoing any study-related activities.
2. Patients with histological documentation of AJCC stage III or IV melanoma of the skin, mucosa, eye or unknown primary.
3. Unable to undergo resection of all metastatic disease.
4. Negative serology for HBV, HCV, HIV and Syphilis. If positive results for HepB or Syphilis indicate immunity and are not indicative of active infection, the patient can enter the study.
5. Adequate venous access that allows to undergo leucapheresis.
6. Having failed first line treatment with DTIC based chemotherapy
7. Full recovery from all prior therapies. A minimum of 4 weeks (6 weeks in case of prior treatment with nitrosurea or Mitomycin C) should separate the last day of prior treatment administration and the date of informed consent.
8. WHO performance status of 0, 1 or 2 (see Appendix D).
9. Male and female patients ≥ 18 years of age.
10. Laboratory parameters should be within normal range, except for the following laboratory parameters, which must be within the ranges specified:see protocol.
11. Viral tests:HIV,HBV and HCV
12. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the study.
13. Patients must be willing to cooperate for the whole period of the study.

Exclusion Criteria:

1. Evidence of immunodeficiency. Autoimmune disease requiring medical treatment
2. Any serious acute or chronic illnesses or other conditions requiring concurrent medications not allowed during this study.
3. History of malignancy.
4. Inability to undergo PET/CT or MRI examination.
5. Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
6. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
7. Subject is pregnant or is currently breast-feeding, anticipates becoming pregnant/ impregnating their partner during the study or within 6 months after study participation, or subject does not agree to follow acceptable methods of birth control, such as hormonal contraception, intra-uterine pessary, condoms or sterilization, to avoid conception during the study and for at least 6 months after receiving the last dose of study treatment.
8. Current alcohol dependence or drug abuse.
9. Known hypersensitivity to the study treatment.
10. Legal incapacity or limited legal capacity.
11. Presence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
12. Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-12; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
a new tumor evaluation (PET/CT) | 24 weeks

SECONDARY OUTCOMES:
Document the anti-melanoma activity | week 8, 16 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Bart Neyns, Professor, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Laken, Brussels Capital, Belgium

REFERENCES:
- [Derived] Wilgenhof S, Van Nuffel AMT, Benteyn D, Corthals J, Aerts C, Heirman C, Van Riet I, Bonehill A, Thielemans K, Neyns B. A phase IB study on intravenous synthetic mRNA electroporated dendritic cell immunotherapy in pretreated advanced melanoma patients. Ann Oncol. 2013 Oct;24(10):2686-2693. doi: 10.1093/annonc/mdt245. Epub 2013 Jul 31. PMID 23904461